CLINICAL TRIAL: NCT02958748
Title: Change of Immune Cell of ARDS Patients：an Observational Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Jianfeng Xie, Doctor, Southeast University, China
Other Study IDs: 20161106
Record Dates: First submitted 2016-11-06; First posted 2016-11-08 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Intensive Care Medicine; ARDS
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- ARDS: Patients admitted to ICU with diagnosis of ARDS,which happened in 48hours.
  Interventions: Other: taking blood sample
- Control: Heathy vonlunteers
  Interventions: Other: taking blood sample

INTERVENTIONS:
Other: taking blood sample

SUMMARY:
To evaluate change of different immune cellsduring ARDS and its impact on prognosis.

ELIGIBILITY:
Inclusion Criteria:

①sign on the acknowledged

②Diagnosis with ARDS(The Berlin definition），onset within 48hours

Exclusion Criteria:

①diagnosis of hematological or immunological disease

②treatment with chemotherapy agents or corticosteroids within 6 months prior to or during the hospitalization.

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Diagnosis:ARDS(The Berlin definition），onset within 48hours Without past history which may impact immune function
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2016-11; Primary Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
mortality | 28-day